CLINICAL TRIAL: NCT06575790
Title: Using Simplified Meal Boluses Versus Carbohydrate Counting in Adolescents With Hybrid Closed Loop Systems: A Randomized Crossover Trial
Brief Title: Using Simplified Meal Boluses Versus Carbohydrate Counting in Adolescents With Hybrid Closed Loop Systems
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24-1159
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple Meal Bolusing (Experimental): Participants will be instructed to enter a set number of carbohydrates before meals based on if they are having a small, medium, or large meal. The preset numbers for meals will be based on their average total daily dose (TDD) determined during the 2-week usual care observation period. The participants will have their insulin to carbohydrate ratios set based on the standard formula of 450/TDD for all meals initially (e.g. a child with a TDD of 50 u/day would have 450/50=9 so an I:C of 1:9). They enter a carbohydrate amount of 30 g for small meals, 60 g for regular meals, and 90 g for large meals.
  Interventions: Behavioral: Simple Meal Bolusing
- Precise Carbohydrate counting (Active Comparator): Participants will be instructed to enter a precise carbohydrate count before meals to the best of their ability. Pump settings may be adjusted per provider discretion and typical clinical care during this time period.
  Interventions: Behavioral: Carbohydrate counting

INTERVENTIONS:
Behavioral: Simple Meal Bolusing — Participants will enter pre-determined numbers for small, medium, or large carbohydrate meals rather than using precise carbohydrate counting
  Arms: Simple Meal Bolusing
Behavioral: Carbohydrate counting — Participants will be instructed to enter accurate carbohydrate counts to the best of their ability for all meals and snacks
  Arms: Precise Carbohydrate counting

SUMMARY:
The goal of this trial is to evaluate blood sugar control in patients with type 1 diabetes when using a simple meal bolus strategy (small, medium, large meals) compared to carbohydrate counting when on a hybrid closed loop system. The main question it aims to answer are:

What is the blood sugar time in range when using simple meal boluses versus carbohydrate counting?

Participants will:

Use the simple meal bolus plan for 4 weeks. Do precise carbohydrate counting for 4 weeks. Provide their continuous glucose monitor and pump data Take surveys about the experience of meal bolusing during the study

DETAILED DESCRIPTION:
This is a prospective randomized crossover trial in adolescents and adults on HCL systems at the Barbara Davis Center for Childhood Diabetes (BDC) with the objective of testing a new simple meal bolus strategy that would not require carbohydrate counting. Given the clear benefit of HCL systems on glycemic control, the ability to use an alternative meal bolus strategy may make HCL systems more accessible. This is a fixed dose of insulin given at meals for small, medium, or large meals that would eliminate the need for precise carbohydrate counting and increase access to patients with low numeracy or difficulty with carbohydrate counting. Although HCL systems cannot yet provide automatic meal bolus insulin, such systems can minimize hyperglycemia through basal modulation and automated correction dosing and should be able to mitigate some of the impact of non-precise carbohydrate coverage. The systems can also help prevent hypoglycemia through basal modulation and pausing insulin delivery. This study will evaluate glycemic control while using the simple meal bolus strategy as compared to traditional precise carbohydrate counting in addition to assessing feasibility, acceptability, and impact on meal-related diabetes burden of each meal bolus strategy.

The proposed study will be a prospective, randomized crossover trial at a single site. Study participants will be randomized via REDCap 1:1 to Group A or Group B with plan for up to a max of 60 total participants to account for drop-out. Neither the participants nor the investigators will be blinded to group assignments due to the nature of the study.

After enrollment, groups will have a 2-week run-in period of usual care. At the first study visit, patients will upload their pump/CGM data, take pre-study surveys, and review carbohydrate counting or simple meal boluses. Pump settings may be adjusted per provider discretion and typical clinical care. Both groups will be instructed to use their systems as they typically would for 4 weeks with the exception of what is entered for carbohydrates for meal boluses. Group B will enter the precise carbohydrate count to the best of their ability, while the Group A will be instructed to enter an assigned number of carbohydrates based on if the meal is small, medium, or large. Participants will have a follow-up visit (in-person, virtual, or by phone) after 4 weeks to provide pump and CGM data, adjust insulin dosing as needed, and review the new strategy. They will have 1 week of usual care as a wash-out period followed by 4 weeks using the opposite strategy. Participants will have a final study visit to upload data and take post-study surveys.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of T1D of at least 1 year duration
* Using a commercial HCL system
* Willingness to not start any new non-insulin glucose-lowering agent during trial
* Willingness to participate in all study procedures
* Investigator has confidence that participant can successfully operate all study devices and adhere to protocol

Exclusion Criteria:

* History of >1 severe hypoglycemic event with seizure or loss of consciousness in the last 6 months or >1 DKA event in the last 6 months not related to illness or infusion set failure
* History of chronic renal disease or currently on hemodialysis, adrenal insufficiency, hypothyroidism that is not adequately treated, use of oral or injectable steroids within the last 8 weeks, or known ongoing adhesive intolerance
* A condition, which in the opinion of the investigator or designee, would put the participant or study at risk
* Participation in another interventional trial at the time of enrollment
* Pregnancy

Ages: 14 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Time in Range | Measured during the duration of the study period, up to 12 weeks
  % of time sensor glucose values are between 70-180 mg/dL

SECONDARY OUTCOMES:
Hypoglycemia | Measured during the duration of the study period, up to 12 weeks
  Percentage of time with BG <70 mg/dL and <54 mg/dL as reported by CGM
Hyperglycemia | Measured during the duration of the study period, up to 12 weeks
  Percentage of time with BG >250 mg/dL as reported by CGM
Feasibility, acceptability, and self-reported mealtime insulin bolus burden | Given 3 times during the duration of the study period, up to 12 weeks
  Survey completed by participants to report on feasibility, acceptability, and self-reported mealtime insulin bolus burden using the different mealtime bolus strategies

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Davis Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No